CLINICAL TRIAL: NCT02376322
Title: A Phase II Trial of Hypofractionated Radiotherapy (16 Gy in 2 Fractions With an Interval of One Week) for the Palliation of Complicated Bone Metastases in Patients With Poor Performance Status
Brief Title: Hypofractionated Radiotherapy (16/2) for the Palliation of Complicated Bone Metastases in Patients With KPS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santa Casa de Porto Alegre (Other)
Responsible Party: Principal Investigator, Mauricio F Silva, Medical Doctor at Radiation Oncology Unity, Santa Casa de Porto Alegre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISCMPA01
Record Dates: First submitted 2015-02-10; First posted 2015-03-03 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Bone Metastases
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: Radiotherapy
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiotherapy in bone metastases (Experimental): The purpose of this one armed, phase II trial is to determine the efficacy and safety profile of a hypofractionated radiotherapy regimen, 16 Gy in 2 fractions with an interval of one week, for the palliation of complicated bone metastases in patients with poor performance status.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Hypofractionated radiotherapy regimen, 16 Gy in 2 fractions in complicated bone metastases in patients with poor performance status

SUMMARY:
Literature has shown that hypofractionated radiotherapy regimens are efficacious in patients with complicated bone metastases and have a low potential for severe treatment-related toxicities. There is a clear need for hypofractionated schedules in the complicated bone metastases population, especially when considering the overarching aim of palliative radiotherapy and the clinical features of this patient population. As well, current research examining hypofractionated approaches in bone metastases patients with impending or pathologic fractures, neuropathic pain or accompanying soft tissue masses has been markedly scarce.

DETAILED DESCRIPTION:
In response the the already commented on, the purpose of this one armed, phase II trial is to determine the efficacy and safety profile of a hypofractionated radiotherapy regimen, 16 Gy in 2 fractions with an interval of one week, for the palliation of complicated bone metastases in patients with poor performance status.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven malignancy.
2. Patients aged 18 and above.
3. Advanced cancer patients with at least one complicated bone metastasis. A complicated bone metastasis will be operationally defined as a bone metastasis that has an accompanying: soft tissue mass or extraosseous component penetrating the normal cortical boundary; neuropathic pain; post surgical intervention for bone fixation; impending fracture or high fracture risk in weight bearing long bone as defined by Harrington's criteria but not surgical candidate: lytic bone lesion involving more than ½ the diameter of the bone cortex , greater than 2.5 cm in greatest diameter, or in the intertrochanteric line (29).
4. Patients with Karnofsky Performance Status (KPS) 30-60 at the time of baseline evaluation.
5. Patients who are planned to receive radiation treatment to the complicated site(s) being followed for study.
6. Patients who had surgery for complicated bone metastases.
7. Patients who are currently taking any systemic therapy (i.e. chemotherapy, hormone therapy, or bone modifying agents) or planning to begin systemic therapy within two weeks of treatment will be allowed to participate in the study; study personnel will note any use of systemic therapy in the study records.
8. Patients who are able to provide a worst pain score at the complicated site(s) being followed for study.
9. Patients who are able and willing to fill out a daily diary.
10. Patients who are able to provide informed consent prior to being enrolled to the study.

Exclusion Criteria:

1. Patients with leukemia or Hodgkin's/non-Hodgkin's lymphoma.
2. Patients who are surgical candidates with pathologic fractures or lesions at high risk for pathologic fracture in the humerus, radius, ulna, femur, tibia, or fibula. They will be eligible for post-operative hypofractionated radiotherapy.
3. Patients with spinal cord compression or cauda equina syndrome.
4. Patients who are currently receiving any radiopharmaceuticals.
5. Patients who are unable to record a pain score, complete a daily diary or to communicate requested information to study personnel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07-30 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
Overall pain response at the site of treatment, which will be measured at two months post-treatment. Pain response will be measured using the International Consensus on Palliative Radiotherapy Endpoints Pain Response Categories. | 2 months after the end of the second radiotherapy fraction
  The general follow up will finish 1 year after each patient inclusion

SECONDARY OUTCOMES:
Quality of life as assessed by the EORTC QLQ PAL-15 and EORTC QLQ-BM22 | General follow up will be 1 year after each patient inclusion
  Quality of life assessed by these 2 questionnaries will follow composite information
Side effects of Radiotherapy. | General follow up will be 1 year after each patient inclusion
  Nausea and vomiting, pain flare, skin rash, esophagitis, mucositis, diarrhea, spinal cord/cauda equina compression, pathologic fracture, re-irradiation rate).

CONTACTS AND LOCATIONS:
Overall Officials: Maurício F Silva, PhD, Principal Investigator — Medical Doctor at Radiation Oncology Unit
Locations (4):
- Brazil (2):
  - ISCMPA, Porto Alegre, Rio Grande do Sul
  - ICESP, São Paulo, São Paulo
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada
- S. Maria Hospital, Terni, Italy